CLINICAL TRIAL: NCT07099053
Title: Amyloid PET Imaging in the Baltimore Longitudinal Study of Aging (BLSA)
Brief Title: Amyloid PET Imaging in the Baltimore Longitudinal Study of Aging
Status: Not yet recruiting | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002099; 002099-AG
Record Dates: First submitted 2025-07-31; First posted 2025-08-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-07-23

CONDITIONS: Aging
Keywords: Amyloid; PET
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults aged 55 and older.: Adults aged 55 and older.

SUMMARY:
Background:

Some people experience cognitive decline as they age. That is, they lose memory, problem-solving, and other mental abilities. Amyloids are groups of proteins that develop in the brain and increase in number as people age. Researchers want to use imaging scans to track amyloids in people s brains over time. Their goal is to find out if any changes are related to cognitive decline or other medical issues.

Objective:

To learn how amyloids may affect brain structure and function as people age.

Eligibility:

People aged 55 years and older who are enrolled in the Baltimore Longitudinal Study of Aging.

Design:

Participants will have imaging scans and other tests every 1 to 4 years, depending on their age. Those 80 and older will be scanned yearly. These scans will be done during regular BLSA visits.

The scans will be positron emission tomography and computed tomography (PET CT). Participants will be given fluid through a tube inserted into a vein in their arm. The fluid is a tracer that will cause the amyloids to light up in the images. Then they will lie on a bed with their head inside a PET CT scanner. They will lie still for about 30 minutes.

Participants will have tests to assess their memory and other mental skills. They will answer questions about their mood and daily life. These tests will take about 40 minutes to complete; they may be done in person or by phone.

Participants will give a contact number for someone who can answer questions about the participant s daily routine. These questions may be answered in person or by phone.

Participants will be in this study for 5 years....

DETAILED DESCRIPTION:
Abstract

We are examining changes in brain structure, function, and neuropathology as predictors of cognitive decline and impairment through longitudinal neuroimaging assessments of selected Baltimore Longitudinal Study of Aging (BLSA) participants at the National Institute on Aging (NIA). The hypothesis driving this study is that accelerated preclinical changes in brain structure and function in specific regions, including mesial temporal cortex, cingulate cortex, precuneus, and inferior parietal cortex, will predict which individuals subsequently develop cognitive impairment and Alzheimer s disease. Since 2005, we have performed serial positron emission tomography (PET) with the radiotracer (11C) Pittsburgh compound B (PiB) to measure amyloid pathology in a subset of participants from the BLSA to investigate the neuropathological basis of memory change and cognitive impairment. Through the protocol we are continuing longitudinal amyloid PET imaging of older participants and evaluating new participants. In conjunction with each BLSA visit, we will perform a single PET scan of (18F) florbetaben (trade name Neuraceq TM) to measure in vivo amyloid distribution in individuals aged 55 years and older. Approximately half of the neuroimaging study participants are enrolled in the BLSA autopsy program, and the integration of autopsy and imaging findings is an active area of investigation to gain a better understanding of factors that promote cognitive resilience in individuals who have amyloid pathology but do not show memory impairment. In addition, we are using neuroimaging tools to investigate modulators of cognitive and brain changes, including sex differences in brain aging, genetic risk factors, and the effects of sex steroid and other hormones. An understanding of these brain-behavior associations and early detection of accelerated brain changes that predict cognitive decline and impairment will be critical in identifying individuals likely to benefit from new interventions.

Objectives:

The principal goal of the project is the acquisition of longitudinal data on regional brain amyloid levels in BLSA participants to investigate these changes in relation to other medical, brain imaging, psychological, and cognitive data collected through the BLSA. Specifically, the primary objectives are to continue to address the following questions:

* What are the rates and regional distribution of changes in brain amyloid pathology in nondemented men and women throughout adulthood?
* What is the frequency and progression of brain amyloid pathology in older adults and what is the clinical significance of these findings for cognitive aging?
* Against a background of age-related changes in brain structure and function, which changes predict cognitive impairment and dementia and when do these changes occur in relation to the onset of amyloid accumulation?
* What factors modulate cognitive and brain aging and how do they impact the relation between amyloid pathology and cognitive outcomes?
* How well do blood-based biomarkers of Alzheimer s disease, collected through the main BLSA study, reflect amyloid pathology in the brain?

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA:
* Participants are men and women 55 years and older drawn from the BLSA sample and thus, represent the gender/ethnic characteristics of this study group. Enrollment is defined as the initial imaging session of the planned longitudinal study.
* Inclusion criteria: BLSA participants who do not meet exclusion criteria and have had or agreed to have an MRI under the BLSA study.
* Participants who lack capacity to consent will not be enrolled in the study. If the participant loses capacity to consent over the course of follow-up they will be removed them from the study. Competency to consent is assessed as part of the BLSA visit and we will not include people who are not competent to provide consent.

EXCLUSION CRITERIA:

* Preexisting central nervous system diseases
* Weight over 300 lbs.
* Active metastatic cancer (except basal cell cancer)
* Implanted electronic hearing devices
* Breast Cancer with radiation treatment
* Lymphoma
* Pacemaker
* Brain tumor
* Shrapnel
* Schizophrenia
* Bipolar disorder
* Epilepsy
* Language barrier that makes it difficult to understand participant.
* Aneurisms greater than 3mm
* Aneurysm clips
* Parkinson s disease/PD medications
* Huntington s disease
* Severe Endocrinopathy- treated thyroid conditions ok; treated, controlled diabetes ok. (exclude HbA1c over 8 which is poorly controlled diabetes)
* Diagnosis of dementia or mild cognitive impairment
* Younger than 55 years of age
* Pregnancy
* Ineligible for MRI
* History of stroke or documented TIAs requiring hospitalization
* Known brain vascular malformations or adenomas
* History of significant radiation exposure
* Those with a Blessed score of 4 or more with the BLSA will be reviewed at a research diagnostic case conference to rule out dementia diagnoses prior to enrollment.

Ages: 55 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women over age 55.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2029-12-12 (Estimated); Study Completion 2029-12-12 (Estimated)

PRIMARY OUTCOMES:
Amyloid accumulation | longitudinal
  yearly PET scans

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Ferrucci, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States